CLINICAL TRIAL: NCT01670019
Title: A Randomized, Blinded, Comparison of Asenapine and Placebo as Adjunctive Treatment in Patients With Non-Psychotic Major Depressive Disorder Incompletely Responsive to Antidepressant Monotherapy
Brief Title: Antidepressant Plus Asenapine Versus Antidepressant Plus Placebo for Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00037462
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Results first posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-08

CONDITIONS: Major Depressive Disorder Without Psychotic Features
Keywords: Depression; Antidepressant; Antipsychotic
MeSH Terms: conditions — Depression | interventions — asenapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asenapine 5-20 mg daily (Experimental): Asenapine will be started at 5 mg BID. The asenapine dose can be increased to 15 mg daily and then to 20 mg daily, or reduced to 5 mg daily, depending on therapeutic response and tolerability
  Interventions: Drug: Asenapine 5-20 mg daily
- Placebo 1-4 tablets daily (Placebo Comparator): Matched, blinded placebo tablets will be administered at doses from 1-4 tablets daily depending on therapeutic response and tolerability
  Interventions: Drug: Placebo 1-4 tablets daily

INTERVENTIONS:
Drug: Asenapine 5-20 mg daily — 5 mg QHS, or 5 mg BID, or 5 mg QAM and 10 mg QHS, or 10 mg BID
  Other Names: SAPHRIS
  Arms: Asenapine 5-20 mg daily
Drug: Placebo 1-4 tablets daily — One placebo tablet QHS, or one placebo tablet BID, or one placebo tablet QAM and two placebo tablets QHS, or two placebo tablets BID
  Other Names: Placebo
  Arms: Placebo 1-4 tablets daily

SUMMARY:
This is a 6-week comparison of asenapine versus placebo as an add-on to ongoing antidepressant treatment in patients with major depression who have not had a complete therapeutic response to treatment with the antidepressant alone.

The investigators hypothesize that added asenapine will produce greater reductions in depression than will added placebo.

DETAILED DESCRIPTION:
The investigators will undertake a 6-week, double-blind, randomized, parallel-group, placebo-controlled trial of adjunctive asenapine in 130 patients with MDD without psychosis who have had an incomplete therapeutic response to treatment with an antidepressant medication alone.

ELIGIBILITY:
Inclusion Criteria:

-130 male or female patients, 18-65 years of age, with:

1. DSM-IV diagnosis of MDD without psychosis (single episode or recurrent) confirmed by the Mini-International Neuro-psychiatric Interview (MINI)
2. MADRS total score > 20, and item 1 (Apparent Sadness) score > 2 at enrollment and randomization
3. Inadequate therapeutic response during their current depressive episode; an inadequate therapeutic response will be defined as continued depressive psychopathology (see criterion 2) following > six weeks of therapy at adequate doses (according to the US label) of any non-tricyclic, non-MAOI antidepressant medication

Exclusion Criteria:

1. Additional DSM-IV Axis I diagnoses other than Generalized Anxiety Disorder, Panic Disorder with or without Agoraphobia, or Social Phobia within 6 months prior to enrollment
2. DSM-IV Axis II diagnoses that significantly impact the current psychiatric status
3. Current MDD episode lasting > 12 months
4. Electroconvulsive therapy within the preceding 6 months
5. Substance or alcohol dependence, as defined by DSM-IV criteria, within 6 months prior to enrollment
6. Unstable medical illness, epilepsy, traumatic brain injury, Parkinson disease, or dementia (MMSE <24)
7. Risk of suicide as defined by MADRS item 10 score > 4
8. Prior failure to respond to asenapine
9. Pregnancy or failure to use an acceptable form of birth control. Pregnancy as determined by serum pregnancy test at baseline
10. Hepatic impairment and history of low WBC, by medical history and interview.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Beyer, MD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - Georgia Health Sciences University, Augusta, Georgia
  - Carolina Behavioral Care, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Brody School of Medicine at East Carolina University, Greenville, North Carolina
  - North Carolina Psychiatric Research Center, Raleigh, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Asenapine 5-20 mg Daily | Placebo 1-4 Tablets Daily
Started | 23 | 23
Completed | 14 | 23
Not Completed | 9 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Asenapine 5-20 mg Daily | Placebo 1-4 Tablets Daily | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.39 (11.34) | 45.87 (12.016) | 45.13 (11.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in MADRS Total Score
Description: The Montgomery Asberg Depression Rating Scale (MADRS) is used by clinicians to assess the severity of depression among patients with a diagnosis of depression. It is designed to be sensitive to change resulting from antidepressant therapy.
  MADRS is a 10-item scale. Each MADRS item is rated on a 0 to 6 scale. The MADRS Total score ranges from 0 (min) to 60 (max). Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Baseline, 6 weeks
Population: Analysis includes those participants who completed week 6 assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Asenapine 5-20 mg Daily | Placebo 1-4 Tablets Daily
Number analyzed (Participants) | 14 | 23
units on a scale | -14.29 (9.73) | -11.61 (11.82)

2. Secondary Outcome: Study Completion Rate
Description: The percentage of patients completing the study in their assigned treatment arm (asenapine or placebo) at the end of 6 weeks
Time Frame: 6 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Asenapine 5-20 mg Daily | Placebo 1-4 Tablets Daily
Number analyzed (Participants) | 23 | 23
percentage of participants | 60.87 | 100

3. Secondary Outcome: Clinical Response Rate
Description: Clinical Response rate will be defined as the number of participants with a > 50% reduction from baseline in MADRS total score.
  MADRS is a 10-item scale. Each MADRS item is rated on a 0 to 6 scale. The MADRS Total score ranges from 0 (min) to 60 (max). Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: Baseline, 6 weeks
Measure: Number; unit: participants
Arm/Group | Asenapine 5-20 mg Daily | Placebo 1-4 Tablets Daily
Number analyzed (Participants) | 14 | 23
participants | 7 | 12

4. Secondary Outcome: Clinical Remission Rate
Description: Clinical Remission will be defined as the number of participants with a MADRS total score < 7.
  MADRS is a 10-item scale. Each MADRS item is rated on a 0 to 6 scale. The MADRS Total score ranges from 0 (min) to 60 (max). Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Asenapine 5-20 mg Daily | Placebo 1-4 Tablets Daily
Number analyzed (Participants) | 14 | 23
participants | 5 | 5

5. Secondary Outcome: Rates of Sustained Remission
Description: Sustained remission will be defined as at least two consecutive post-randomization assessments (weeks 2, 4, and 6) during which minimal depressive psychopathology (MADRS < 7) is present.
  MADRS is a 10-item scale. Each MADRS item is rated on a 0 to 6 scale. The MADRS Total score ranges from 0 (min) to 60 (max). Higher MADRS scores indicate higher levels of depressive symptoms.
Time Frame: 2, 4, 6 weeks
Population: Participants that completed all data collection timepoints at week 2, 4, 6.
Measure: Number; unit: participants
Arm/Group | Asenapine 5-20 mg Daily | Placebo 1-4 Tablets Daily
Number analyzed (Participants) | 13 | 23
participants | 4 | 4

ADVERSE EVENTS:
Arm/Group | Asenapine 5-20 mg Daily | Placebo 1-4 Tablets Daily
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 16/23 | 16/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Asenapine 5-20 mg Daily (N=23) | Placebo 1-4 Tablets Daily (N=23)
Insomnia (Psychiatric disorders) | 11 | 11
Excessive daytime sedation (Psychiatric disorders) | 10 | 12
Oral/ Lingual dysaethesia (Gastrointestinal disorders) | 5 | 2
orthostasis faintness (Nervous system disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No